CLINICAL TRIAL: NCT07362108
Title: Cardiovascular Events Related to the Coronary Artery Treated by Surgical or Percutaneous Revascularization in Patients With Stable Multivessel Coronary Artery Disease: A Long-Term Comparison With Medical Therapy - Target Trial
Brief Title: Cardiovascular Events Related to Treated Coronary Arteries in Stable Multivessel CAD
Status: Completed | Type: Observational
Sponsor: Instituto do Coracao (Other Government)
Responsible Party: Principal Investigator, Thiago Ovanessian Hueb, MD, PhD, Instituto do Coracao
Other Study IDs: SDC 6147 25 158
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease; Stable Coronary Artery Disease; Multivessel Coronary Artery Disease; Myocardial Ischemia
Keywords: Coronary artery bypass grafting; Percutaneous coronary intervention; Medical therapy; Stable coronary artery disease; Multivessel disease; Vessel-related outcomes; Myocardial infarction; Cardiac death; MASS study
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Myocardial Infarction; Death | interventions — Coronary Artery Bypass; Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Coronary Artery Bypass Grafting (CABG): Patients with stable multivessel coronary artery disease treated with surgical coronary artery bypass grafting.
  Interventions: Procedure: Coronary Artery Bypass Grafting
- Percutaneous Coronary Intervention (PCI): Patients with stable multivessel coronary artery disease treated with percutaneous coronary intervention.
  Interventions: Procedure: Percutaneous Coronary Intervention
- Medical Therapy: Patients with stable multivessel coronary artery disease treated exclusively with optimized medical therapy.
  Interventions: Other: Optimized Medical Therapy

INTERVENTIONS:
Procedure: Coronary Artery Bypass Grafting — Surgical myocardial revascularization using coronary artery bypass grafting.
  Groups: Coronary Artery Bypass Grafting (CABG)
Procedure: Percutaneous Coronary Intervention — Percutaneous coronary intervention performed according to standard clinical practice.
  Groups: Percutaneous Coronary Intervention (PCI)
Other: Optimized Medical Therapy — Guideline-directed medical therapy for stable coronary artery disease.
  Groups: Medical Therapy

SUMMARY:
This retrospective cohort study evaluates cardiovascular events directly related to treated coronary arteries in patients with stable multivessel coronary artery disease. Outcomes in patients undergoing coronary artery bypass grafting or percutaneous coronary intervention will be compared with those receiving optimized medical therapy alone. This study aims to improve understanding of how different treatment strategies impact long-term vessel-related outcomes in patients with stable multivessel coronary artery disease.

DETAILED DESCRIPTION:
Previous studies evaluating coronary revascularization strategies have relied on broad composite endpoints, which may include events unrelated to the treated vessel. This study focuses on vessel-related outcomes, specifically non-fatal myocardial infarction and cardiac death attributable to the treated coronary artery. Patients were selected from the MASS (Medicine, Angioplasty, or Surgery Study) database at a single tertiary center. By analyzing vessel-specific events, this study aims to provide a more accurate assessment of the long-term impact of different treatment strategies in stable multivessel coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable multivessel coronary artery disease, defined as ≥70% stenosis in at least two major epicardial coronary arteries, with documented myocardial ischemia and clinical indication for surgical, percutaneous, or medical treatment.

Exclusion Criteria:

* Patients with limited life expectancy, severe left ventricular dysfunction (ejection fraction <35%), recent acute coronary syndrome, recent revascularization procedures, significant valvular disease, chronic kidney disease (creatinine ≥2.0 mg/dL), active malignancy, or inability to complete long-term follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with stable multivessel coronary artery disease and documented myocardial ischemia, selected from the MASS (Medicine, Angioplasty, or Surgery Study) database at a single tertiary academic center.
Sampling Method: Non-Probability Sample
Enrollment: 1695 (Actual)
Dates: Start 1995-01-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Non-fatal myocardial infarction related to the treated coronary artery | Up to 5 years of follow-up
Cardiac death attributable to the treated coronary artery | Up to 5 years of follow-up

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly because this study is based on a retrospective institutional database with data ownership governed by institutional policies and local data protection regulations. De-identified data may be made available upon reasonable request, subject to approval by the investigators and the institutional ethics committee.